CLINICAL TRIAL: NCT06105606
Title: Feasibility of the AveCure Microwave Ablation Technology for the Bronchoscopic Treatment of Malignant Central Airway Obstructions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: MedWaves, Inc (Unknown)
Responsible Party: Principal Investigator, Jason A Beattie, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-131
Record Dates: First submitted 2023-07-05; First posted 2023-10-27 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Airway Obstruction; Central Airway Obstruction
Keywords: Endoluminal malignant central airway obstruction; Central airway obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- AvuCure Microwave Ablation (Experimental): Participants will undergo study procedures as follows:
  * Baseline assessments
  * Hospital admission for bronchoscopy under general anesthesia and microwave ablation via standard of care.
  * Participants will be followed at 1, 3, and 6 months post-procedure.
  Interventions: Device: AveCure Flexible Microwave Ablation Probe

INTERVENTIONS:
Device: AveCure Flexible Microwave Ablation Probe — Consists of a handheld, surgical device which delivers microwave energy from its microwave antenna. The flexible probe has a 3cm active microwave field that radiates from the tip.
  Other Names: Avecure 16 Gauge Probe Model 16-123-01-15

SUMMARY:
This research is being done to evaluate the feasibility of the AveCure Flexible Microwave destruction of tissue (Ablation) Probe for the treatment of malignant central airway obstruction using a thin, tube-like instrument with a light and a lens for viewing and removing tissue (bronchoscopic).

The name of the intervention being used in this research study is:

AveCure Flexible Microwave Ablation Probe (handheld, surgical device that delivers microwave energy via flexible probe tip)

DETAILED DESCRIPTION:
This research study is a prospective, single-arm, cohort study to evaluate the feasibility of Microwave Ablation (MWA) Probe for the bronchoscopic treatment of malignant lesions causing central airway obstructions (COA). The AveCure prob will be placed in contact with the COA to treat with energy.

The U.S. Food and Drug Administration (FDA) has approved this intervention for use throughout the body, but it has not been approved for the specific indication of central airway obstruction.

Research study procedures include screening for eligibility, hospitalization for bronchoscopy and MWA, blood tests, survey questionnaires, Computerized Tomography (CT) scan imaging, and pulmonary function tests.

Participation in this research study is expected to last about 6 months.

It is expected that about 10 people will take part in this research study.

MedWaves, Inc is funding this research study by providing the ablation probe and generator.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 18 and 80 years of age and able to provide informed consent.
* Candidate for bronchoscopy under general anesthesia.
* Diagnosis of central airway obstruction (trachea, right main stem bronchus, left main stem bronchus), as evidenced by CT or CT/PET imaging confirmed or suspected to be due to malignant etiology, for which the bronchoscopist has deemed that endoscopic ablation/debridement is indicated (i.e. endobronchial tumors, mixed endobronchial/extrinsic compression lesions).

Exclusion Criteria:

* Patients who are unable to understand the informed consent, including potential risks and benefits of the procedure.
* Patients in whom bronchoscopy under general anesthesia is contraindicated.
* Any comorbidity that the investigator feels would interfere with the safety of the subject or the evaluation of study objectives
* Pacemaker, implantable cardioverter, or another electronic implantable device
* Patients with coagulopathy
* Patients in other therapeutic lung cancer studies
* COVID-19 positive patient at the time of the procedure.
* Patients who are pregnant
* Patients with purely extrinsic compression of the airway.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Failure Rate (FFR) | 6 months
  Feasibility of the AveCure microwave technology to ablate a target malignant central and lobar airway lesions causing > 50% obstruction, defined as at least 9/10 of the planned ablations (90%) successfully performed bronchoscopically according to the study protocol

SECONDARY OUTCOMES:
6-month airway patency rate | 6 months
  6-month airway patency rate defined as the proportion of participants achieve airway patency. Airway patency will be calculated as the minimal airway luminal area at the CAO as a percentage of the average of the distal and proximal airway luminal areas.
Grade 3-5 Treatment-related Toxicity Rate | Adverse events evaluated 1, 3 and 6 month after procedure.
  All grade 3-5 adverse events (AE) with attribution of possibly, probably or definitely related to neoadjuvant treatment based on CTCAEv5 are counted. Rate is the proportion of treated participants with at least one post-baseline safety assessment experiencing at least one of these adverse events during the time of observation.
Airway Obstruction (AO) Rate | CT scan at 1, 3, 6 and 12 months after procedure
  AO Rate defined as percentage of airway obstruction assessed at bronchoscopy and on CT scan after the study procedure measured through the Myer-Cotton grading system and percentage change in luminal cross sectional area. Central airway obstruction (CAO) is defined as occlusion of more than 50% of the trachea, mainstem bronchi, bronchus intermedius, or a lobar bronchus.
Change in Subjective Perception of Dyspnea | Assessed 1, 3, 6 and 12 months after procedure.
  subjective perception of dyspnea as measured by the modified Medical Research Council dyspnea scale (mMRC)
Number and type of additional tools that are used during bronchoscopy. | Index procedure only (at ablation).
Procedural Bleeding | Index procedure only (at ablation).
  bleeding assessed by the Nashville scale
Change in peak flow measurement | Baseline to 30 days +/- 7 days post ablation
  Peak flow measurement using a standard peak flow meter will also be performed by research staff.
6-month Overall Survival (OS) | 6 months
  6-month OS is a probability estimated using the Kaplan-Meier method; OS is defined as the time from study entry to death, or censored at date last known alive.
6-month mechanical ventilation-free survival | 6 months
  6-month mechanical ventilation-free survival is a probability estimated using the Kaplan Meier method; PFS is defined as the duration of time from study entry to documented mechanical ventilation.
Histologic characteristics of tissue ablated with the AveCure microwave technology device. | Index procedure only (at ablation).
MW number of energy applications | Index procedure only (at ablation)
MW time of application | Index procedure only (at ablation)
  seconds
Total time of MW ablation | Index procedure only (at ablation)
  seconds
Total energy delivered during MW ablation | Index procedure only (at ablation)
  mW
Temperature during ablation | Index procedure only (at ablation)
  degrees Celsius
Length of ablation procedure | Index procedure only (at ablation)
  minutes
Change in Quality of Life (QoL) as measured by Saint George Respiratory Questionnaire (SGRQ) | ssessed 1, 3, 6 and 12 months after procedure.
Procedural bleeding | Index procedure only (at ablation)
  estimated blood loss (mL)
Change in Quality of Life (QoL) measured by European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ-C30) | Assessed 1, 3, 6 and 12 months after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Beattie, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu